CLINICAL TRIAL: NCT03003455
Title: Nasotracheal Intubation Over a Bougie Placed Via a Subsequently Removed Nasal Trumpet
Brief Title: Nasotracheal Intubation Over a Bougie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Abrons, Ron O, Assistant Professor of Anesthesiology, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201112757
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Nasotracheal Intubation; Nasal Bleeding
Keywords: Nasotracheal Intubation
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Nasotracheal Intubation (CVT) (Active Comparator): Blind passage of an endotracheal tube via the nare followed by videolaryngoscopy-assisted passage through the glottis, with or without the aid of Magill forceps
  Interventions: Procedure: Conventional Nasotracheal Intubation
- Nasotracheal Intubation Over a Bougie (NIB) (Experimental): Nasotracheal intubation over a bougie, placed with videolaryngoscopy assistance, via a nasopharyngeal airway with or without the aid of Magill forceps
  Interventions: Procedure: Nasotracheal intubation over a bougie

INTERVENTIONS:
Procedure: Nasotracheal intubation over a bougie — Nasotracheal intubation over a bougie, placed with videolaryngoscopy assistance, via a nasopharyngeal airway with or without the aid of Magill forceps
  Other Names: Abrons technique for nasotracheal intubation; Nasotracheal intubation over a bougie placed via a subsequently removed nasal trumpet; NIB
  Arms: Nasotracheal Intubation Over a Bougie (NIB)
Procedure: Conventional Nasotracheal Intubation — Blind passage of an endotracheal tube via the nare followed by videolaryngoscopy-assisted passage through the glottis, with or without the aid of Magill forceps
  Other Names: CVT
  Arms: Conventional Nasotracheal Intubation (CVT)

SUMMARY:
The purpose of this study is to determine whether nasal intubation over a bougie placed via a nasal trumpet will decrease nasal trauma when compared to the conventional technique of blind nasal endotracheal tube passage.

DETAILED DESCRIPTION:
Conventional nasotracheal intubation techniques (or "Conventional Videolaryngoscopic Techniques," CVT) are known to be associated with significant trauma to the patient's nares and the endotracheal tube itself. The investigators propose an alternative technique (Nasotracheal intubation over a bougie placed via a subsequently removed nasal trumpet, or NIB) which involves using Seldinger technique over a bougie placed via a nasal trumpet which promises to not only be less traumatic to the patient and the endotracheal tube, but also to take less time to perform and have a higher first-attempt success rate than conventional methods. The investigators propose a randomized prospective interventional study comparing this new technique with conventional technique to see if a significant difference exists.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery with an anesthetic plan including asleep nasotracheal intubation

Exclusion Criteria:

* Patients needing emergent airway protection
* Patients undergoing emergency surgery
* Patients whom are known to be pregnant
* Patients whom are currently anticoagulated (including daily aspirin use)
* Patients whose anesthetic includes the use of nitrous oxide
* Patients whom are currently incarcerated
* Patients 7 years of age or younger
* Mentally incompetent adults
* Patients whom refuse involvement in the study

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2012-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Nasal trauma | 60-90 seconds post-intubation
  Bleeding noted on nasopharyngeal exam by surgical resident

SECONDARY OUTCOMES:
Nasal trauma | 5 minutes post-intubation
  Bleeding noted on nasopharyngeal exam by surgical resident
Time to intubation | Measured immediately post-intubation
  Time from first entrance of ETT or bougie into the nare to the presence of end-tidal CO2 via nasotracheal ETT
First attempt success rate | Measured immediately post-intubation
  Whether or not there was successful nasotracheal intubation on the first attempt
Need for Magill forceps | Measured Immediately post-intubation
  Whether or not Magill forceps were used during airway management

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elwood T, Stillions DM, Woo DW, Bradford HM, Ramamoorthy C. Nasotracheal intubation: a randomized trial of two methods. Anesthesiology. 2002 Jan;96(1):51-3. doi: 10.1097/00000542-200201000-00014. PMID 11753001
- [Background] O'Connell JE, Stevenson DS, Stokes MA. Pathological changes associated with short-term nasal intubation. Anaesthesia. 1996 Apr;51(4):347-50. doi: 10.1111/j.1365-2044.1996.tb07746.x. PMID 8686823
- [Background] Morimoto Y, Sugimura M, Hirose Y, Taki K, Niwa H. Nasotracheal intubation under curve-tipped suction catheter guidance reduces epistaxis. Can J Anaesth. 2006 Mar;53(3):295-8. doi: 10.1007/BF03022218. PMID 16527796
- [Background] Abrons RO, Vansickle RA, Ouanes JP. Seldinger technique for nasal intubation: a case series. J Clin Anesth. 2016 Nov;34:609-11. doi: 10.1016/j.jclinane.2016.06.027. Epub 2016 Jul 19. PMID 27687457
- [Background] Cossham PS. Nasotracheal tube placement over a bougie. Anaesthesia. 1997 Feb;52(2):184-5. No abstract available. PMID 9059115